CLINICAL TRIAL: NCT07120984
Title: A Phase II Study to Evaluate the Safety and Efficacy of L19TNF With Alkylating Chemotherapy for Patients With Recurrent IDH-mutant Astrocytoma or Oligodendroglioma
Brief Title: A Study to Evaluate the Safety and Efficacy of L19TNF With Alkylating Chemotherapy for Patients With Recurrent IDH-mutant Astrocytoma or Oligodendroglioma
Acronym: IMAGLIO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFGLIO-02/25
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Temozolomide; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1: perioperative cohort of patients with recurrent astrocytoma or oligodendroglioma (Experimental): patients will be treated with 1 cycle (D1, D3 and D5) L19TNF before resection and 4 weeks after surgery
  Interventions: Biological: L19TNF
- 2A:L19TNF Monotherapy for patients with recurrent oligodendroglioma (Experimental): patients with IDH-mutant oligodendroglioma, WHO Grade 2 or 3 at first progression after radiotherapy and one line of systemic chemotherapy, are treated with up to 6 cycles of 6 weeks with L19TNF
  Interventions: Biological: L19TNF monothery in recurrent oligodendroglioma
- 2B1: L19TNF plus TMZ for patients with recurrent oligodendroglioma (Experimental): patients with IDH-mutant oligodendroglioma, WHO Grade 2 or 3 at first progression after radiotherapy and one line of systemic CCNU-based chemotherapy, are treated with L19TNF and temozolomide chemotherapy TMZ
  Interventions: Biological: L19TNF and TMZ
- 2B2: L19TNF plus CCNU for patients with recurrent oligodendroglioma (Experimental): patients with IDH-mutant oligodendroglioma, WHO Grade 2 or 3 at first progression after radiotherapy and one line of systemic temozolomide chemotherapy, are treated with L19TNF and CCNU
  Interventions: Biological: L19TNF and CCNU
- 3A: L19TNF monotherapy for patients with recurrent astrocytoma (Experimental): patients with IDH-mutant astrocytoma, WHO Grade 2, 3 or 4 at first progression after radiotherapy and one line of systemic chemotherapy, are treated with L19TNF
  Interventions: Biological: L19TNF monotherapy
- 3B1: L19TNF plus TMZ for patients with recurrent astrocytoma (Experimental): patients with IDH-mutant astrocytoma, WHO Grade 2, 3 or 4 at first progression after radiotherapy and one line of systemic CCNU-based chemotherapy, are treated with L19TNF and temozolomide chemotherapy TMZ
  Interventions: Biological: L19TNF and TMZ in recurrent astrocytoma
- 3B2: L19TNF plus CCNU for patients with recurrent astrocytoma (Experimental): patients with IDH-mutant astrocytoma, WHO Grade 2, 3 and 4 at first progression after radiotherapy and one line of systemic chemotherapy including temozolomide, are treated with L19TNFand CCNU
  Interventions: Biological: L19TNF and CCNU in recurrent astrocytoma

INTERVENTIONS:
Biological: L19TNF — 1 cycle of TNF before resection and 6 cycles after surgery
  Arms: 1: perioperative cohort of patients with recurrent astrocytoma or oligodendroglioma
Biological: L19TNF and TMZ — 6 cycles of 28 days with L19TNF and TMZ
  Arms: 2B1: L19TNF plus TMZ for patients with recurrent oligodendroglioma
Biological: L19TNF and CCNU — 6 cycles of 6 weeks of L19TNF and CCNU every 6 weeks
  Arms: 2B2: L19TNF plus CCNU for patients with recurrent oligodendroglioma
Biological: L19TNF monotherapy — 6 cycles of 6 weeks with L19TNF
  Arms: 3A: L19TNF monotherapy for patients with recurrent astrocytoma
Biological: L19TNF and TMZ in recurrent astrocytoma — 6 cycles of 28 days with L19TNF (D1, D3, D5) and temozolomide chemotherapy TMZ (D1-5).
  Arms: 3B1: L19TNF plus TMZ for patients with recurrent astrocytoma
Biological: L19TNF and CCNU in recurrent astrocytoma — 6 cycles of 6 weeks of L19TNF (D1, D3, D5, D22, D24 and D26) and CCNU (D1) every 6 weeks
  Arms: 3B2: L19TNF plus CCNU for patients with recurrent astrocytoma
Biological: L19TNF monothery in recurrent oligodendroglioma — 6 cycles of 6 weeks with L19TNF
  Arms: 2A:L19TNF Monotherapy for patients with recurrent oligodendroglioma

SUMMARY:
The purpose of this study is to explore the safety and efficacy of the antibody-cytokine fusion protein L19TNF alone or in combination with alkylating chemotherapy in patients with recurrent IDH mutant glioma.

DETAILED DESCRIPTION:
This protocol describes an open label, multi-centric phase 2 study and patients will be treated with L19TNF at 13µg/kg as monotherapy or in combination with alkylating chemotherapy (Lomustine or Temozolamide) in different cohorts:

* COHORT 1: L19TNF monotherapy in perioperative cohort of patients with recurrent astrocytoma or oligodendroglioma,
* COHORT 2A: L19TNF Monotherapy for patients with recurrent oligodendroglioma,
* COHORT 2B1: L19TNF plus TMZ for patients with recurrent oligodendroglioma,
* COHORT 2B2: L9TNF plus CCNU for patients with recurrent oligodendroglioma,
* COHORT 3A: L19TNF Monotherpay for patients with recurrent astrocytoma,
* COHORT 3B1: L19TNF plus TMZ for patients with recurrent astrocytoma,
* COHORT 3B2: L19TNF plus CCNU for patients with recurrent astrocytoma.

Eligibility criteria in this trial are:

* Age ≥18
* IDH-mutant glioma at first recurrence or progression after alkylating chemotherapy:
* COHORT 1: Grade ≥2 oligodendroglioma or astrocytoma with planned resection
* COHORT 2A, 2B1, 2B2: Grade ≥2 oligodendroglioma
* COHORT 3A, 3B1, 3B2: Grade ≥2 astrocytoma
* No therapy for first recurrence or progression after alkylating chemotherapy, except resection.
* Patients must have measurable disease according to RANO 2.0
* Karnofsky Performance Status (KPS) ≥ 70%.

The primary endpoint of the study is the Progression Free Survival Rate at 12 months (PFS-12).

The following secondary endpoints are considered:

* Progression-free survival (PFS)
* Overall response rate (ORR)
* Disease control rate
* Duration of response (DoR)
* Overall survival (OS)
* Safety and tolerability: adverse event (AE), serious AE (SAE), Drug-induced liver injury (DILI), physical examinations, echocardiography, ECG and standard laboratory parameters (hematology, biochemistry liver and urine analysis)
* Human anti-factor antibodies (HAFA)
* popPK

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. IDH-mutant glioma (according to WHO 2021 classification) at first recurrence or progression after alkylating chemotherapy:

   * COHORT 1: Grade ≥2 oligodendroglioma or astrocytoma with planned resection, tumor tissue from prior resection must be available
   * COHORT 2A: Grade ≥2 oligodendroglioma
   * COHORT 2B1: Grade ≥2 oligodendroglioma previously treated with lomustine as monotherapy or in combination
   * COHORT 2B2: Grade ≥2 oligodendroglioma previously treated with temozolomide as monotherapy or in combination
   * COHORT 3A: Grade ≥2 astrocytoma
   * COHORT 3B1: Grade ≥2 astrocytoma previously treated with lomustine as monotherapy or in combination
   * COHORT 3B2: Grade ≥2 astrocytoma previously treated with temozolomide as monotherapy or in combination
3. Measurable disease according to RANO 2.0 criteria.
4. Documented IDH1 and/or IDH2 gene mutations detected by immunochemistry or sequencing.
5. Karnofsky Performance Status (KPS) ≥ 70%.
6. Life expectancy ≥ 3 months.
7. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV, negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
8. Female patients: female patients must be either documented not Women Of Childbearing Potential (WOCBP)* or must have a negative pregnancy test within 14 days of starting treatment. Additionally WOCBP must agree to use, from the screening to 6 months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.

   Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required from the screening to 6 months following the last administration of temozolomide, lomustine or L19TNF.
9. Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Any therapy for recurrence/progression after alkylating chemotherapy, except resection.
2. Therapy for glioma within 4 weeks of start of study treatment.
3. Surgical resection of glioma within 4 weeks of start of study treatment.
4. Stereotactic biopsy of glioma within 2 weeks of start of study treatment.
5. Inability to undergo contrast-enhanced MRI.
6. Known history of allergy to TNF or lomustine or temozolomide, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
7. Absolute neutrophil count (ANC) < 1.5 x 10^9/L; platelets < 100 x 10^9/L or hemoglobin (Hb) < 9.0 g/dl.
8. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min/1.73m2 or for patients older than 65 years without albuminuria or proteinuria, creatinine clearance < 45 mL/min/1.73m2.
9. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 1.5 x ULN).
10. INR > 1.5 ULN.
11. Any severe concomitant condition, which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
12. Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent, in the judgement of the investigator.
13. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
14. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
15. Clinically significant cardiac arrhythmias or requiring permanent medication.
16. LVEF < 55% or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered clinically significant by the investigator. Patients with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of QTc >470 milliseconds using Fredricia's QT correction formula) are excluded.
17. Uncontrolled hypertension, defined by systolic blood pressure ≥ 140 mmHg and diastolic blood pressure ≥ 90 mmHg.
18. Arterial aneurism at high risk of rupture.
19. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
20. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders.
21. Anxiety ≥ CTCAE Grade 3.
22. Severe diabetic retinopathy, such as severe non-proliferative retinopathy and proliferative retinopathy.
23. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
24. Known history of tuberculosis.
25. Pregnancy or breast feeding.
26. Requirement of chronic administration of high dose steroids or other immunosuppressant drugs. Subjects must have been either off steroids, or on a stable or decreasing dose ≤ 4 mg daily dexamethasone (or equivalent) for 7 days prior to start of treatment. Limited or occasional use of steroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
27. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
28. Concurrent malignancies other than glioma unless the patient has been disease-free without intervention for at least 2 years.
29. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
30. Serious, non-healing wound, ulcer or bone fracture.
31. Deep vein thrombosis, pulmonary embolism or other acute vascular events within 6 months.
32. Anticoagulation therapy with P2Y12 antagonists (e.g., clopidogrel, ticagrelor) and vitamin K antagonists (e.g., phenprocoumon, warfarin).
33. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
34. Any live vaccination within 4 weeks prior to treatment or plan to receive live vaccination during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | The PFS rate will be assessed at 12 months (PFS-12) in IDH mutant astrocytoma and in oligodendroglioma.
  Progression-free survival (PFS) in according to RECIST v.1.1. The duration is defined beginning from randomization to progression or death from any cause.

IPD SHARING:
Plan to Share IPD: No